CLINICAL TRIAL: NCT03956420
Title: ERAS Implementation in Coronary Artery Bypass Surgery
Brief Title: Enhanced Recovery After Surgery (ERAS) in Coronary Artery Bypass Graft / Off Pump Coronary Artery Bypass (CABG/OPCAB)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Ewa Kucewicz-Czech, Clinical Professor, Head of Unit, Silesian University of Medicine
Other Study IDs: KNW/0022/KB1/26/18
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Coronary Artery Bypass Surgery/Grafting, ERAS
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Preoperative Period; Postoperative Period; Intraoperative Period

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Implemented ERAS (Early Recovery After Surgery) elements
  Interventions: Behavioral: Premedication visit; Dietary Supplement: Preoperative period; Drug: Preoperative period; Other: Postoperative period; Other: Intraoperative period; Drug: Intraoperative period
- Control group: The control group will consist of patients treated during the study in accordance with the current standards used in the Department

INTERVENTIONS:
Behavioral: Premedication visit — detailed information about surgery, anaesthesia and postoperative period
  Groups: Study group
Dietary Supplement: Preoperative period — avoidance of prolonged fasting, intake of fluids with carbohydrates before surgery
  Groups: Study group
Drug: Preoperative period — administration of melatonin 5 mg in the evening and pregabalin 75 mg one hour before entering the operating theatre
  Groups: Study group
Other: Postoperative period — Fluids 1 ml/kg/h; Discontinuation of propofol at the moment of drainage and cardiovascular system stabilization; Fluids administered orally 2 hours after extubation; Early mobilisation
  Groups: Study group
Other: Intraoperative period — deep temperature (necessity to maintain normothermia during the stay in the operating theatre 36 °C. Normothermia should be maintained rather than restored.
  Other Names: Normothermia
  Groups: Study group
Drug: Intraoperative period — Pyralgin 1 g i.v. after induction of anaesthesia; in patients allergic to Pyralginum, Perfalgan 1 g i.v.
  Groups: Study group
Drug: Intraoperative period — Ketamine 30 mg i.v. after induction of anaesthesia
  Groups: Study group
Drug: Intraoperative period — Sevoflurane 1.5 MAC higher in patients < 60 years old
  Groups: Study group
Drug: Intraoperative period — Propofol infusion in patients at risk of postoperative vomiting (Apfel ≥ 2 points), sevoflurane administration at the moments of strong stimuli from the operating field
  Groups: Study group
Drug: Intraoperative period — Continuous infusion of balanced multi-electrolyte fluids 1-3 ml/kg/h
  Groups: Study group

SUMMARY:
It has been assumed that some elements of the ERAS protocol may contribute to the reduction of complications and improve the satisfaction of patients undergoing coronary artery bypass surgery.

Elements of the ERAS strategy will be tested in this study. The elements that prove to be feasible and have a positive effect on the treatment process will be introduced into everyday clinical practice.

In the next stage of the research, we are planning to investigate whether the introduction of the ERAS strategy has had a long-term positive effect on the quality of life after treatment (a survey 1 month and 6 months after leaving the hospital).

DETAILED DESCRIPTION:
Evaluation of the impact of implemented elements of the ERAS strategy on the results of surgical treatment of coronary artery disease in the aspect of:

* preoperative preparation (comprehensive information, premedication, hydration),
* haemodynamic stability (discontinuation of angiotensin-converting enzyme inhibitors and angiotensin II receptor blockers immediately before surgery), optimal pre- and intraoperative fluid therapy,
* occurrence of respiratory complications (assessment of the duration of mechanical ventilation and passive oxygen therapy),
* demand for painkillers in the postoperative period, after introducing the preemptive strategy,
* incidence of postoperative delirium,
* time to recovery of the normal bowel function (nausea, vomiting),
* possibility of early mobilisation on the first day after surgery,
* patient's satisfaction with treatment assessed on the basis of a survey carried out on the day before leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

* CABG/OPCAB (Coronary Artery Bypass Surgery/Off Pump Coronary Bypass Surgery).
* Left ventricular ejection fraction above 35% (EF ≥ 35%).
* The operation was performed in a planned mode.

Exclusion Criteria:

* Haematological diseases and the associated increased risk of bleeding in the early postoperative period. Patients taking anticoagulants until the day of surgery with the exception of aspirin.
* Neurological disorders, stroke with persistent symptoms, dementia.
* Chronic lung disease with hypoxia and the need for regular medication.
* Inability to move independently, disability preventing efficient rehabilitation, prolonged use of painkillers.
* Emergency surgery, reoperation.
* Return to the operating room regardless of the reason (resternotomy).
* Perioperative infarction with circulatory destabilization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet the inclusion criteria will be eligible for the study. The perioperative period and anaesthesia will be supervised by anaesthesiologists trained to carry out the study. The study group will include 50 patients. The results obtained in the study group will be compared with the results of the control group. The control group will consist of patients treated during the study in accordance with the current standards used in the Department.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
ERAS bundle compliance in the first 72 hours post-op | 72 hours post operation
  Number of interventions for the ERAS protocol that are delivered to patient (numeric data e.g. 5 out of 10)
Shorter Length Of Hospitalization (LOH) | up to 4 weeks after operation
  Total amount of days spent in hospital

SECONDARY OUTCOMES:
Preoperative anxiety | on admission to the operating unit
  Assessment of patient's emotional status according to Anxiety Likert Scale (consisted of five evenly spaced numbers each anchored to a level of anxiety: 1="not at all anxious," 2="a little anxious," 3="moderately anxious," 4="very anxious," 5="extremely anxious)
Time to extubation | 0 -72 hours
  Time taken until patient extubated post operation (in hours)
Assessment of postoperative pain | 0-24 hours
  Pain scores at 6hours, Numeric scale 0 (no pain) - 10 (severe pain)
Incidence of postoperative nausea and vomiting | At moment 0, 3, 6, 12 and 24 hours after extubation
  To calculate the PONV Impact Scale score, add the numerical responses to questions 1 and 2. A PONV Impact Scale score of ≥5 defines clinically important PONV (Q1. Have you vomited: 0. No
  1. Once
  2. Twice
  3. Three or more times Q2. Have you experienced a feeling of nausea :0. Not at all
  1. Sometimes 2. Often or most of the time 3. All of the time)
Time to drink | 0-72 hours
  Time until patient first drinks post extubation (in hours)
Time to eating | 0-72 hours
  Time until patient first eats post extubation (in hours)
Time to bowel movement | in hours after extubation, up to 1 week
  Hours elapsed to event
Incidence of postoperative delirium | in hours after extubation, up to 72 hours
  Delirium Screening according to Nursing Delirium Screening Scale, Each feature is scored on 0-2 based on severity, with 0=absent, 1=mild, and 2=severe.
  Positive Nu-DESC is score ≥2, maximum total score is 10
Postoperative complications | up to 2 weeks after surgery
  Rate measurement
Time to mobilisation | 0-72 hours
  First mobilisation with nurse/physiotherapist post-op (in hours)

OTHER OUTCOMES:
Quality of Recovery | 1 and 6 months after operation
  This process resulted in the QoR-15 questionnaire ( Part A: How have you been feeling in the last 24 hours; 0-10 0-poor, 10 - excellent; rated areas: breath,food,feeling rested, sleep, hygiene,communicate, getting support, return to work, feeling comfortable, well-being; Part B Have you had any of following in the last 24h: modreate pain, severe pain, nause or vomiting, feeling worried, feeling sad; 10-0, 10 - none of the time, 0 - all of the time

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Kucewicz-Czech, Study Chair — Upper-Silesian Medical Centre; DEPARTMENT OF ANAESTHESIOLOGY AND INTENSIVE CARE WITH CARDIAC MONITORING
Locations (1):
- Upper-Silesian Medical Centre of the Silesian Medical University, Katowice, Polska, Poland

IPD SHARING:
Plan to Share IPD: No